CLINICAL TRIAL: NCT00006166
Title: The North American Study for the Treatment of Refractory Ascites (NASTRA) Clinical Trial
Brief Title: North American Study for the Treatment of Refractory Ascites (NASTRA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NASTRA (completed); 1R01DK051523 (NIH)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Ascites; Liver Cirrhosis
Keywords: refractory ascites; paracenteses
MeSH Terms: conditions — Ascites; Liver Cirrhosis

INTERVENTIONS:
Procedure: Transjugular intrahepatic portasystemic shunts (TIPS)
Procedure: Total paracentecis (TP)

SUMMARY:
The NASTRA Clinical Trial is a multi-center, randomized, controlled clinical trial designed to determine if treatment with transjugular intrahepatic portasystemic shunts (TIPS) is superior to high volume paracentesis (total paracentesis, TP) for the treatment of refractory ascites due to cirrhosis. Only patients with clinically tense symptomatic ascites (shortness of breath, umbilical hernia, abdominal pain and/or distension, and/or limitation of activity) who have either diuretic-resistant ascites or diuretic-intractable ascites are being studied.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis as documented by biopsy or clinical/laboratory parameters WITH
* Tense symptomatic ascites and need for paracentesis (10 L) within last 2 months AND
* Failure of medical therapy as defined by the inability to lose at least 3.3 lbs/week while on maximum doses of diuretics or diuretic related complications (severe hyponatremia, hypercalcemia, azotemia or encephalopathy)

Exclusion Criteria:

* Causes of ascites other than cirrhosis and portal hypertension
* Terminal liver failure
* Portal vein thrombosis
* Congestive heart failure
* Acute renal failure
* Active encephalopathy
* Alcoholic hepatitis
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-03; Study Completion 2001-10

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - University of Miami Hospital, Miami, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oregon Health Sciences University, Portland, Oregon
  - Medical College of Virginia Hospitals, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- The Toronto Hospital, Toronto, Ontario, Canada